CLINICAL TRIAL: NCT06143722
Title: Camrelizumab Plus Chemotherapy in Combination With Synchronous or Sequential Radiotherapy for Advanced Esophageal Squamous Cell Carcinoma With Oligometastases: a Randomized Controlled Phase II Clinical Study
Brief Title: Synchronous or Sequential Radiotherapy for Advanced Esophageal Squamous Cell Carcinoma With Oligometastases.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ting Liu, Clinical Investigator, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WestChinaHS
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Advanced Esophageal Squamous Carcinoma With Oligometastases
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: A randomized, prospective phase II trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous radiotherapy group (Experimental)
  Interventions: Radiation: simultaneous with radiotherapy
- Sequential radiotherapy group (Active Comparator)
  Interventions: Radiation: synchronous with radiotherapy

INTERVENTIONS:
Radiation: simultaneous with radiotherapy — Chemotherapy combined with immunotherapy simultaneous with radiotherapy
  Arms: Simultaneous radiotherapy group
Radiation: synchronous with radiotherapy — Chemotherapy combined with immunotherapy synchronous with radiotherapy
  Arms: Sequential radiotherapy group

SUMMARY:
A randomized, prospective phase II trial was conducted to explore the timing of radiotherapy intervention in combination with chemotherapy and immunotherap in order to provide an effective treatment for patients with advanced esophageal squamous carcinoma with oligometastases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old, male or female;
* Patients with pathologically diagnosed esophageal squamous cell carcinoma;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and <10% weight loss within six months;
* Patients with distant organ metastasis or nonregional lymph node metastasis, or distant organ/nonregional lymph node metastasis with regional lymph node metastasis, as defined by the AJCC 8th edition;
* All positive regional lymph nodes were counted as one lesion, and adjacent metastatic nonregional lymph nodes could be treated as one lesion;
* All metastases must be amenable to local radiotherapy;
* 5 or fewer metastatic lesions including tumor beds and recurrent anastomoses, ≤ 4 metastatic lesions in any organ system, and a maximum lesion diameter ≤ 5 cm;
* not including fading lesions during prior therapy (i.e., no longer visible on CT or metabolically active eliminated on PET-CT);
* All metastases have not received local treatment such as radiotherapy, surgery, radiofrequency ablation prior to enrollment (Lesions located in the area of prior radiotherapy may be considered target lesions if progression is confirmed and considered measurable according to RECIST 1.1);
* Measurable lesions ≥1 cm (maximum diameter) determined by CT or MRI, or ≥2 cm by other radiologic techniques, according to RECIST criteria;
* Expected survival time of at least 12 weeks;
* No previous surgery, chemotherapy, radiation therapy or immunotherapy for any cancer within the past 6 months;
* Laboratory test indicators meet the following criteria:

  ①Bone marrow function: hemoglobin (Hb) ≥80g/L; white blood cell count (WBC) ≥lower limit of normal; absolute neutrophil count (ANC) ≥1.5×10^9 /L; platelet count ≥80×109 /L;

  ②Renal function: Cr ≤ ULN (upper limit of normal) × 1.5, endogenous creatinine clearance (Ccr) ≥ 45 ml/min;

  ③Liver function: total bilirubin ≤ ULN × 1.5; ALT and AST ≤ ULN × 2.5; (if there is liver metastasis, total bilirubin is not higher than 3 times the upper limit of normal, and transaminases are not higher than 5 times the upper limit of normal);

  ④Coagulation function: international normalized ratio of prothrombin time ≤ ULN × 1.5, and partial thromboplastin time within the normal value;
* Females of child-bearing potential agree to use contraception during the study period and for 6 months after the completion of the study; patients who have had a negative serum or urine pregnancy test within seven days prior to enrollment in the study and who are not breastfeeding; and males agreeing to use contraception during the study period and for 6 months after the completion of the study;
* Subjects who can understand the study situation and voluntarily sign the informed consent form;
* Patients are expected to be compliant and able to follow up on efficacy and adverse events according to protocol requirements.

Exclusion Criteria:

* Metastases with faint borders making radiotherapy treatment infeasible; metastases located within 3 cm of previously irradiated structures;
* Poor nutritional status with a BMI < 18.5 Kg/m^2, if symptomatic nutritional support was corrected prior to randomization to group, enrollment may be considered after evaluation by the principal investigator;
* Severe impairment of lung function.
* patients with an esophageal mediastinal fistula and/or esophagotracheal fistula prior to treatment or at risk of invasion of vital vessels with lethal bleeding;
* Diagnosis of other malignant tumors (except carcinoma in situ, basal cell carcinoma, etc.) within the previous 5 years;
* Presence of any active autoimmune disease or history of autoimmune disease; immunodeficiency, active tuberculosis, hepatitis B ( hepatitis B virus titer HBV-DNA <500 IU/ml after treatment and if liver function is normal will be allowed), or positive test for hepatitis C virus.
* Presence of hereditary or acquired bleeding and thrombotic tendencies;
* Treatment with immunosuppressive drugs or corticosteroids (> 10 mg prednisone or equivalent per day) within 14 days prior to enrollment; patients are allowed to receive steroid therapy to control CNS-related symptoms, but the dose must ≤ 5 mg per day of dexamethasone (or equivalent); in the absence of an active autoimmune disease, inhaled or topical steroids and adrenal gland replacement dosing are acceptable; alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are permitted; patients with experimental medications that require premedication with corticosteroids are not restricted;
* Allergic reaction to any of the study drugs or contraindication to radiotherapy;
* Participation in another clinical trial within 30 days prior to enrollment;
* Individuals considered by the investigator to be unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 12 months
  Progression-free survival will be measured as time to either progression or death.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 months
  Overall survival will be measured as time to death from any cause.
Disease Control Rate (DCR) | 12 months
  The DCR was defined as the proportion of patients with the best efficacy (complete response or partial response or stable disease).
Objective response rate (ORR) | 12 months
  Defined as the response to treatment as assessed by the investigator based on the Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) criteria, containing cases of complete response, and partial response.
Adverse events | 12 months.
  toxicity values caused by treatment.